CLINICAL TRIAL: NCT00659581
Title: Special Survey (Survey on Cerebrovascular and Cardiovascular Events Under Long-term Use) of Micardis Tablets (Telmisartan)
Brief Title: J-TARGET,Japanese Telmisartan Study for Antihypertensive Good Effect in Long Term Observation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.511
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertension
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan — Oral administration

SUMMARY:
The primary objective of this post marketing survey is to prospectively investigate patients with hypertension treated with Micardis Tablets (hereinafter "this drug") in routine clinical settings for 3 years in order to determine the following:

1. Adverse events and adverse drug reactions under long-term use
2. Blood pressure measurements during the survey period
3. Determination of the incidence of cerebrovascular and cardiovascular events under use of this drug in routine clinical settings
4. Patient's lifestyle and background factors that are considered to affect the occurrence of cerebrovascular and cardiovascular events

ELIGIBILITY:
Inclusion criteria:

Hypertension patients unadministered Micardis.

Exclusion criteria:

1. Patients with a history of hypersensitivity to any ingredient of this product.
2. Pregnant woman or possibly pregnant woman
3. Patients with extremely poor bile secretion or patients with serious hepatic disorder

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese hypertension patients
Sampling Method: Probability Sample
Enrollment: 21471 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the survey, 21,433 patients were enrolled. The data of 439 patients have not reported after the registration, and 551 patients were not observed after the registration: 38 entry violation, 24 contract violation, 493 no office visit after initial prescription and 9 undefined study medication (the numbers were overlapping).
Period: Overall Study
Arm/Group | Telmisartan
Started | 20994
Completed | 12412
Not Completed | 8582
Not completed — Adverse Event | 1006
Not completed — Lack of Efficacy | 1183
Not completed — Other | 6393

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan
Number analyzed (Participants) | 20443
Age, Continuous [Mean (Standard Deviation); unit: years old] | 64.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10278
  Male | 10165

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cerebrovascular(CeV) and Cardiovascular (CaV) Events
Time Frame: 3 years after initiation of treatment
Population: All of observed 20,443 patients were included as intention to treat set
Measure: Number; unit: Number of participants
Arm/Group | Telmisartan
Number analyzed (Participants) | 20443
Number of participants
  Number of patients with CeV and CaV events | 479
  Number of patients with no CeV and CaV events | 19964

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at 6 Months
Time Frame: initiation and 6 months
Population: The 2503 patients with insufficient study medication adherence, no measured systolic blood pressure in the period, or discontinued before 6 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 17940
mmHg | -20.6 (19.9)

3. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at 6 Months
Time Frame: initiation and 6 months
Population: The 2506 patients with insufficient study medication adherence, no measured diastolic blood pressure in the period, or discontinued before 6 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 17937
mmHg | -10.3 (12.5)

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at 12 Months
Time Frame: initiation and 12 months
Population: The 4400 patients with insufficient study medication adherence, no measured systolic blood pressure in the period, or discontinued before 12 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 16043
mmHg | -22.2 (19.9)

5. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at 12 Months
Time Frame: initiation and 12 months
Population: The 4400 patients with insufficient study medication adherence, no measured diastolic blood pressure in the period, or discontinued before 12 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 16043
mmHg | -11.3 (12.8)

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at 24 Months
Time Frame: initiation and 24 months
Population: The 6544 patients with insufficient study medication adherence, no measured systolic blood pressure in the period, or discontinued before 24 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 13899
mmHg | -23.9 (20.2)

7. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at 24 Months
Time Frame: initiation and 24 months
Population: The 6544 patients with insufficient study medication adherence, no measured diastolic blood pressure in the period, or discontinued before 24 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 13899
mmHg | -12.3 (12.8)

8. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at 36 Months
Time Frame: initiation and 36 months
Population: The 8267 patients with insufficient study medication adherence, no measured systolic blood pressure in the period, or discontinued before 36 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 12176
mmHg | -25.0 (19.9)

9. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at 36 Months
Time Frame: initiation and 36 months
Population: The 8270 patients with insufficient study medication adherence, no measured diastolic blood pressure in the period, or discontinued before 36 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan
Number analyzed (Participants) | 12173
mmHg | -13.1 (13.0)

ADVERSE EVENTS:
Time Frame: From signing the informed consent through the end of study
Arm/Group | Telmisartan
Serious Adverse Events (participants affected / at risk) | 1058/20443
Other Adverse Events (participants affected / at risk) | 0/20443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan (N=20443)
Anaemia (Blood and lymphatic system disorders) | 3
Aplastic anaemia (Blood and lymphatic system disorders) | 2
Blood disorder (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Erythropenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 12
Angina pectoris (Cardiac disorders) | 90
Angina unstable (Cardiac disorders) | 3
Aortic valve disease mixed (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 8
Atrioventricular block complete (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 76
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 5
Cardiac sarcoidosis (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 58
Myocardial ischaemia (Cardiac disorders) | 1
Myocardial rupture (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 2
Sick sinus syndrome (Cardiac disorders) | 3
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 3
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Primary hyperaldosteronism (Endocrine disorders) | 1
Cataract (Eye disorders) | 3
Retinal detachment (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 3
Colitis ischaemic (Gastrointestinal disorders) | 2
Colitis ulcerative (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 5
Diverticular perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 5
Intestinal obstruction (Gastrointestinal disorders) | 4
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mesenteric occlusion (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 3
Rectal lesion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 1
Death (General disorders) | 35
Drowning (General disorders) | 1
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 3
Multi-organ failure (General disorders) | 2
Oedema peripheral (General disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 4
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 4
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 3
Appendicitis (Infections and infestations) | 1
Arteriosclerotic gangrene (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Dacryocystitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 2
Gallbladder abscess (Infections and infestations) | 1
Gangrene (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Meningitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Peritoneal tuberculosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 16
Pneumonia bacterial (Infections and infestations) | 11
Pneumonia fungal (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pulmonary tuberculoma (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Pyometra (Infections and infestations) | 1
Sepsis (Infections and infestations) | 9
Septic shock (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Accident (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 11
Femoral neck fracture (Injury, poisoning and procedural complications) | 10
Femur fracture (Injury, poisoning and procedural complications) | 5
Foot fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 5
Head injury (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 1
Internal injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 5
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 6
Uterine rupture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 11
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 16
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adult T-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 42
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 2
Brain stem haemorrhage (Nervous system disorders) | 2
Brain stem infarction (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Cerebellar haemorrhage (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 31
Cerebral infarction (Nervous system disorders) | 169
Convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 6
Dementia Alzheimer's type (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dyskinesia (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Monoplegia (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Quadriplegia (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 13
Transient ischaemic attack (Nervous system disorders) | 22
Vertebral artery stenosis (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 5
Eating disorder (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 4
Diabetic nephropathy (Renal and urinary disorders) | 13
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Lupus nephritis (Renal and urinary disorders) | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Nephropathy (Renal and urinary disorders) | 1
Nephrosclerosis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 4
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 9
Renal failure acute (Renal and urinary disorders) | 4
Renal failure chronic (Renal and urinary disorders) | 23
Renal impairment (Renal and urinary disorders) | 6
Urinary incontinence (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Caplanas syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 9
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aortic anastomosis (Surgical and medical procedures) | 1
Aortic valve replacement (Surgical and medical procedures) | 2
Coronary angioplasty (Surgical and medical procedures) | 1
Dialysis device insertion (Surgical and medical procedures) | 1
Orthopedic procedure (Surgical and medical procedures) | 1
Vascular graft (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 6
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 5
Aortic occlusion (Vascular disorders) | 1
Aortic rupture (Vascular disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Arteriosclerosis obliterans (Vascular disorders) | 7
Blood pressure inadequately controlled (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Intermittent claudication (Vascular disorders) | 2
Shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study is prospective observational study with no limitation of other antihypertensive treatment in compliance with Japanese Pharmaceutical Affairs Law (JPAL) and Good Post-marketing Study Practice (GPSP).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes